CLINICAL TRIAL: NCT07070258
Title: Pediatric Intensive Care Transport Registry
Acronym: PIT Registry
Status: Recruiting | Type: Observational
Sponsor: Philipps University Marburg (Other)
Collaborators: Deutsche Interdisziplinäre Vereinigung für Intensiv- und Notfallmedizin (Other)
Responsible Party: Principal Investigator, Dr. med. Nadine Mand, Head of Neonatology and Pediatric Intensive Care, Department of Pediatrics, Marburg, Philipps University Marburg
Other Study IDs: REG-EK-270072024
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Critical Care Medicine; Transportation of Patients; Pediatrics
Keywords: intensive care transport; critical care transport; pediatrics; registry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill children undergoing interhospital pediatric intensive care transport: All critically ill children undergoing interhospital pediatric intensive care transport, aged at least 27 days and with a corrected gestational age of over 41 weeks, are eligible for inclusion. The upper age limit for enrolment is 18 years. Critical care transports are defined as transports that meet at least one of the following criteria: I) The transport was performed by a dedicated critical care transport team using an intensive care ambulance (Type C vehicle) or an air ambulance. II) The transport was accompanied by a specialist in intensive care or emergency medicine. III) The in-hospital destination of the transport is a critical care area, such as an intensive care unit, a trauma room, a resuscitation area, an operating theatre, an emergency imaging procedure or an emergency intervention.

SUMMARY:
The aim is to establish a nationwide registry for pediatric intensive care transports in Germany. The project aims to describe and analyse the need for, and current practice of, specialised transports. These data could then be used for future demand planning.

DETAILED DESCRIPTION:
In contrast to critical care transport of adults or newborns, transport of pediatric critical care patients in Germany is neither regulated by law nor centrally organized. Due to their different therapeutic needs compared to newborns or adults, critically ill children may receive insufficient treatment during transport. In some regions in Germany, pediatric centers provide specialized pediatric retrieval teams, while others organize each transport individually. Currently, no valid data on pediatric critical care transports in Germany are available, nor are they recorded in a structured manner.

A nationwide registry for pediatric intensive care transports in Germany was initiated to describe and analyze the need for and current practice of these specialized transports.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill children aged at least 27 days and a corrected gestational age of over 41 weeks AND
* Maximum age of 17 years AND
* Interhospital transport AND
* Critical care transport by a dedicated critical care transport team using an intensive care ambulance (Type C vehicle) or an air ambulance OR
* The transport was accompanied by a specialist in intensive care or emergency medicine. OR
* The in-hospital destination of the transport is a critical care area, such as an intensive care unit, a trauma room, a resuscitation area, an operating theatre, an emergency imaging procedure or an emergency intervention.

Ages: 27 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All critically ill children undergoing interhospital pediatric intensive care transport and arriving at a participating center.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Most frequent reason for pediatric intensive care transport | At enrollment

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University of Dresden, Dresden
  - Philipps University of Marburg, Marburg

IPD SHARING:
Plan to Share IPD: No